CLINICAL TRIAL: NCT00105326
Title: A Double-blind, Placebo-controlled, Randomized Study Evaluating the Effect of Paliperidone ER Compared With Placebo on Sleep Architecture in Subjects With Schizophrenia
Brief Title: Trial Evaluating Paliperidone Extended-Release (ER) Tablets Versus Placebo on Sleep in Schizophrenia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002281
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Schizophrenia; Insomnia
Keywords: Schizophrenia; Schizophrenia-related insomnia; insomnia; paliperidone; placebo; polysomnography
MeSH Terms: conditions — Schizophrenia; Sleep Initiation and Maintenance Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: paliperidone ER

SUMMARY:
The primary objective of this study is to evaluate the amelioration of the sleep architecture of patients with schizophrenia and schizophrenia-related insomnia, treated with either 9 mg of extended-release paliperidone ER or placebo, using polysomnography.

DETAILED DESCRIPTION:
Paliperidone is the major active substance produced by the metabolism of risperidone in the body. In patients with schizophrenia, risperidone has been shown to improve the quality of sleep. Therefore it is possible that treatment of paliperidone may improve sleep quality and potentially the quality of life in these patients. The goal of this study is to test the hypothesis that paliperidone improves sleep architecture. This trial is a multicenter, double-blind (neither the patient nor the physician will know if placebo or drug is being given and at what dose), randomized (patients will be assigned to different treatment groups based solely on chance), placebo-controlled study in patients with schizophrenia and schizophrenia related insomnia. The study consists of 2 phases: a screening phase of up to 14 days and a double-blind phase of 15 days. The primary purpose of this study is to evaluate improvement of the sleep architecture of patients with schizophrenia and schizophrenia-related insomnia, treated with either 9 mg/day of paliperidone ER or placebo for 14 days, using polysomnography. In this study, polysomnography (polygraphic recording during sleep of multiple body functions related to the state and stages of sleep to assess possible biological causes of sleep disorders) will be used to measure sleep architecture and continuity. Measurements will be taken on 2 days during the screening phase (averaged for the baseline value) and on the last 2 days of the treatment phase (averaged for the end point value) and will include measurement of non-rapid eye movement (NREM) sleep (including the 4 stages of sleep) and measures of rapid eye movement (REM) sleep. Other assessments pertinent to the continuity and efficiency of sleep such as sleep latency (the length of time that it takes to go from full wakefulness to Stage 2 sleep), sleep efficiency (proportion of sleep during time in bed), sleep maintenance (period of time between sleep onset and awakening and number of awakenings), and sleep duration (total sleep time) will also be measured. At baseline, on Day 7, and at end of treatment, the Positive and Negative Syndrome Scale (PANSS) will be used to assess the symptoms of schizophrenia and the Clinical Global Impression Scale - Severity (CGI-S) will be used to assess the severity of a patients condition. Safety assessments include the incidence of adverse events throughout the study; daily measurement of vital signs (blood pressure, pulse, and temperature); clinical laboratory tests performed both before the study initiation and at end of treatment; and measurement of extrapyramidal symptoms using scales (EPS scales) at baseline, Day 7 and end point. 9 mg of paliperidone ER or placebo taken orally once daily on Days 1 to 14

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia and schizophrenia-related insomnia, no relapse or psychosis for at least 3 months before screening, and considered symptomatically stable
* have apnea/hypopnea score <10 and periodic leg movement score with an arousal index <10
* Weigh >/= 50 kg (>/=110 lbs), with a BMI >/= 18 and </= 35 kg/m2, inclusive
* Agree to adhere to sleep schedule
* Have a sleep history of a minimum of 1.5 hours of wakefulness out of 8 hours in bed.

Exclusion Criteria:

* Current history of suicidal or violent behavior or have exhibited this behavior within the past 6 months
* diagnosis of primary insomnia
* unstable blood pressure
* sleep problems related to general medical conditions, or substance abuse
* diagnosis of or evidence of narcolepsy
* preexisting severe gastrointestinal narrowing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2005-02; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The change from baseline at endpoint in sleep architecture and continuity measurements including sleep time, latency to sleep onset and to persistent sleep, sleep efficiency, time awake & awakenings after sleep onset, Stage 3&4 sleep duration, REM sleep

SECONDARY OUTCOMES:
Changes in the PANSS scores from baseline to end of treatment and the CGI-S score at each time point. Incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Luthringer R, Staner L, Noel N, Muzet M, Gassmann-Mayer C, Talluri K, Cleton A, Eerdekens M, Battisti WP, Palumbo JM. A double-blind, placebo-controlled, randomized study evaluating the effect of paliperidone extended-release tablets on sleep architecture in patients with schizophrenia. Int Clin Psychopharmacol. 2007 Sep;22(5):299-308. doi: 10.1097/YIC.0b013e3281c55f4f. PMID 17690599